CLINICAL TRIAL: NCT02644031
Title: Evaluation of Post-endodontic Pain After Root Canal Treatment With Two Rotary Systems : Mtwo & Safe-sider
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7203
Record Dates: First submitted 2015-12-13; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Pain, Postoperative
Keywords: Instrumentation; Post-operative pain; Root canal preparation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mtwo rotary system (Experimental): ( continuous rotation system)
  Interventions: Procedure: mtwo rotary system
- safe-sider rotary system (Experimental): (reciprocating system)
  Interventions: Procedure: safe-sider rotary system
- hand files (Experimental): k-files
  Interventions: Procedure: hand files

INTERVENTIONS:
Procedure: mtwo rotary system — post-treatment pain after using mtwo rotary system
  Arms: Mtwo rotary system
Procedure: safe-sider rotary system — post-treatment pain after using safe-sider rotary system
  Arms: safe-sider rotary system
Procedure: hand files — post-treatment pain after using hand files
  Arms: hand files

SUMMARY:
Post-endodontic pain (PP) still is major problem for endodontic patients, analgesics are routinely prescribed. Incidence of PP is reported extensively, and reviewed. PP is a complicated multi factorial process and is affected by factors related to patients, to the tooth and to the skills and experience of the dentist and because of that, if the interrelation of these factors is not considered in a PP, study data might be confusing. Any study trying to evaluate the effect of a specific technique or new device in the incidence or characteristics of PP should control all the confounding factors that have been described to be involved in the tested outcome.

reports mention a variable prevalence of PP, ranging from 82.9 to 10.6%. These variations are because of the differences in study methods, and treatment procedures after root canal treatment, selection of patients or experience and skills of the dentists, vary when different studies are compared.

Many studies had confirmed that chemomechanical debridement of the root canal results in extrusion of dentinal chips, pulp tissue fragments, necrotic tissues, microorganisms, and root canal irrigants through the apical foramen. All preparation techniques and instruments, regardless of maintaining shorter working length of the apical terminus have reported to be related with extrusion of infected debris, and some of them extruded less material and others extruded more.

Periapical inflammation and postoperative flare-ups may result from apical extrusion of debris that is also referred to as the "worm" of necrotic debris A common outcome of the studies examining the amount of apically extruded debris was that the techniques involving a push-pull filing motion usually produce a greater mass of apical debris than those have rotational action Files which has reciprocating and in-and-out filing motion, may act as a piston, extruding more debris and irrigants. While the file with continuous rotation motion like a screw conveyor improving transportation of dentinal chips and debris coronally.

In this study, investigators compare post-endodontic pain between these two systems. Mtwo ( continuous rotation system) with safe-sider (reciprocating system). Therefore, the aim of this study is Evaluation of post-endodontic pain after root canal treatment with two rotary systems: Mtwo & safe-sider

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-50 years
* the systemically healthy
* first or second molar teeth require root canal therapy
* irreversible Pulpitis signed without the apical
* root canal curvature of less than 25 degrees, according to Schneider techniques

Exclusion Criteria:

* Root canal treatment,
* history of medication (antibiotics, NSAID, opiates) of the patient 12 hours before treatment ,
* pregnancy,
* complex anatomy,
* channels blocked in the x-ray plate,
* internal and external resorption,
* open apex teeth,
* periodontal disease,
* inflammation and abscesses,
* sinus tract,
* presence of radiographic lesions,
* tooth sensitivity to percussion,
* absence of occlusal contact .

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Information regarding post-operation pain is gathered via a patient using questionnaire and is measured via the visual analogue scale. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: eshaghali saberi, professor, Study Chair — professor of endodontics department
Locations (1):
- Zahedan University of Medical Science, Zahedan, Sistan and Baloochestan, Iran

IPD SHARING:
Plan to Share IPD: Undecided